CLINICAL TRIAL: NCT05783882
Title: Multicenter Open-label Study of the Efficacy, Pharmacokinetica and Safety of Prolgolimab 250 mg Q3W in Patients With Unresectable or Metastatic Melanoma
Brief Title: Prolgolimab 250 mg Q3W in Patients With Unresectable or Metastatic Melanoma
Acronym: FLAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-100-8
Record Dates: First submitted 2023-02-02; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-01

CONDITIONS: Unresectable or Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Prolgolimab

INTERVENTIONS:
Drug: Prolgolimab — 250 mg Q3W

SUMMARY:
Multicentre, single-arm, open-label efficacy, pharmacokinetics, and safety study to demonstrate non-inferiority of prolgolimab 250 mg every 3 weeks versus historical data for prolgolimab 1 mg/kg every 2 weeks in patients with unresectable or metastatic melanoma, as well as collecting pharmacokinetics and safety data.

The study is conducted under the same conditions as the previously conducted study BCD-100-2/MIRACULUM. This means that this Study No. BCD-100-8/FLAT has identical parameters such as:

* selection criteria for subjects in the study, defining the population,
* research centers,
* procedures for evaluating effectiveness and safety,
* permitted prior and concomitant therapy of the underlying disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and the subject's ability to comply with the protocol requirements.
* Age ≥18 years at the time of informed consent.
* Histologically confirmed unresectable or metastatic melanoma (with available documented evidence of relevant examinations).
* Primarily detected advanced or metastatic melanoma, or the disease progression on or after previous systemic therapy.
* Measurable target tumor lesions (at least 1 lesion) according to RECIST 1.1 criteria, confirmed by an independent reviewer.
* ECOG score 0-1.
* Absence of severe organ and system disorders.
* Life expectancy of at least 12 weeks at screening.
* For patients of childbearing potential: willingness to use reliable methods of contraception throughout the study, from the time of informed consent and for up to 6 weeks after the last dose of the study drug.
* Available blocks for a histological examination and/or the patient's consent for collection of biopsy43 samples to obtain histological material to assess the PD-L1 status.

Exclusion Criteria:

* Patients with severe concomitant disorders, life-threatening acute complications of the primary disease (including massive pleural, pericardial, or peritoneal effusions requiring intervention, pulmonary lymphangitis) at the time of informed consent.
* CNS metastases that are progressing or associated with clinical symptoms (e.g., cerebral edema, spinal compression) or requiring the use of glucocorticosteroids and/or anticonvulsants;
* Ongoing concomitant diseases at the time of screening increasing the risk of severe adverse events during the study treatment.
* The need for glucocorticoids or any other drugs with immunosuppressive effects.
* Hematologic abnormalities.
* Renal impairment.
* Hepatic impairment.
* Increased LDH >2 ULN.
* Prior treatment with anti-CTLA4 and/or anti-PD-1/PD-L1/PDL-2 drugs.
* Prior targeted therapy.
* A history of malignancies, except for radically treated diseases in remission for over 5 years prior to starting the study.
* Conditions limiting the patient's ability to comply with the protocol requirements (dementia, neurologic or mental disorders, drug or alcohol addiction, etc).
* Simultaneous participation in other clinical studies55 or participation in other clinical studies within 30 days prior to starting the study treatmen.
* Acute infections or activation of chronic infectious diseases within 28 days prior to the beginning of the study treatment.
* Active hepatitis B, active hepatitis C, HIV-infection, syphilis.
* Impossibility to administer the study drug intravenously.
* Impossibility to perform imaging examinations requiring administration of intravenous contrast media.
* Hypersensitivity to any of the components of BCD-100.
* A history of hypersensitivity to monoclonal antibody products.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 month
  Overall response rate (partial response+complete response rates) according to RECIST 1.1

SECONDARY OUTCOMES:
Overall response rate | 6 month
  Overall response rate (partial response+complete response rates) according to irRECIST
Disease control rate | 6 month
  Disease control rate (stabilization + partial response + complete response rates) according to RECIST 1.1
Disease control rate | 6 month
  Disease control rate (stabilization + partial response + complete response rates) according to irRECIST
Time to response | 6 month
  The time from the frirst administered dose to the response (partial or complete) according to RECIST 1.1
Time to response | 6 month
  The time from the frirst administered dose to the response (partial or complete) according to irRECIST
Duration of Response | 6 month
  Time from the response (partial or complete) repoerted date to the progression or death.

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - State Budgetary Institution of Healthcare of the Arkhangelsk Region "Arkhangelsk Regional Clinical Oncology Dispensary" (SBHI AR ARCOD), Arkhangelsk
  - State Budgetary Institution of Healthcare "Clinical Oncology Dispensary of Chelyabinsk Region" (SBIH CODCR), Chelyabinsk
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - State Budgetary Healthcare Institution "Moscow Clinical Scientific Center funded by Moscow Health Department" (SBHI MCSC MHD), Moscow
  - Federal State Budgetary Institution "N.N. Petrov Research Institute of Oncology" of the Ministry of Healthcare of the Russian Federation, Research Department of the Innovative Methods of Therapeutic Oncology and Rehabilitation, Saint Petersburg
  - Federal State Budgetary Institution "N.N. Petrov Research Institute of Oncology" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tjulandin S, Demidov L, Moiseyenko V, Protsenko S, Semiglazova T, Odintsova S, Zukov R, Lazarev S, Makarova Y, Nechaeva M, Sakaeva D, Andreev A, Tarasova A, Fadeyeva N, Shustova M, Kuryshev I. Novel PD-1 inhibitor prolgolimab: expanding non-resectable/metastatic melanoma therapy choice. Eur J Cancer. 2021 May;149:222-232. doi: 10.1016/j.ejca.2021.02.030. Epub 2021 Apr 17. PMID 33872982